CLINICAL TRIAL: NCT06775951
Title: Appropriateness of Colonoscopy Indication: an Evaluation of the Clinical and Economic Impact. Multicenter Prospective Observational Study.
Brief Title: Appropriateness of Colonoscopy Indication: an Evaluation of the Clinical and Economic Impact.
Acronym: PROMOTE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PROMOTE
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Control and Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection for each patient on endoscopic examination: Data collection in patients undergoing colonoscopy, to identify the ability of the predictive model to predict colonoscopies with significant diagnostic findings, in patients already initiated for diagnostic examination as part of the normal care pathway.

SUMMARY:
The aim of the study is to evaluate the appropriateness of colonoscopy prescription and the impact of colonoscopies in diagnostic performance in order to develop and validate a predictive model for selecting patients most likely to present with significant lesions and thus lower costs and waiting lists.

DETAILED DESCRIPTION:
Colonoscopy is the most frequently conducted endoscopic examination in industrialized countries, occupying a considerable number of personnel and resources. However, colonoscopy is often over-prescribed, resulting in great waste of resources and increased risk to the patient with no discernible benefit. Colonoscopy has many indications and needs precise prescribing criteria to avoid inappropriate use of resources, especially in an open-access health care system such as the Italian one, criteria recently systematized by EPAGE (European Panel for Appropriateness in Gastrointestinal Endoscopy) and ASGE (American Society for Gastrointestinal Endoscopy) based on a set of observational studies. In these studies, it has been shown that colonoscopies with an appropriate indication frequently find significant lesions compared with colonoscopies prescribed according to inappropriate criteria, which are often negative. The aim of the study is to evaluate the appropriateness of colonoscopy prescription and the impact of colonoscopies in diagnostic performance in order to develop and validate a predictive model for selecting patients most likely to present with significant lesions and thus lower costs and waiting lists.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients undergoing outpatient and inpatient colonoscopy for any pathology, as part of the normal care process
* Obtaining informed consent.

Exclusion Criteria:

* Investigations performed in an emergency/emergency setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating subjects will undergo data collection at the same time as colonoscopy. After enrollment, information will be collected for each included patient regarding the demographic and clinical characteristics, the reason for prescription, and the diagnostic question proposed in congruity with EPAGE/ASGE criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1410 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of colonoscopies | 5 months
  Define the number of colonoscopies with indication appropriate out of the total number of colonoscopies performed, and quantify clinically relevant lesions and CCRs in appropriate and inappropriate colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Fuccio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna

IPD SHARING:
Plan to Share IPD: No